CLINICAL TRIAL: NCT06030128
Title: Core Stabilization Exercise Therapy in Chronic Lower Back Pain Management in Community Dwelling Older Adults
Brief Title: Core Stabilization Exercise Therapy in Chronic Lower Back Back Management in Community Dwelling Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Patrick Kwong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230506002
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Low-back Pain; Older Adults; Core Stabilization Exercise Therapy

STUDY DESIGN:
Intervention Model Description: 75 participants will be randomized into the intervention group. Another 75 participants will be randomized into the waiting list control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stabilization exercise group (Experimental): All participants will undergo 16 session exercise program for 2 months. Each session will last for 60minutes. The exercise program will be arranged in a group format with class size ranging from 6 - 8per class. Subjects will be divided into experimental and control groups.
  Interventions: Behavioral: core stabilization exercise
- waiting list control group (No Intervention): Participants in the control group will not receive exercise training at first but were evaluated at the same time as participants in the experimental group.

INTERVENTIONS:
Behavioral: core stabilization exercise — All participants will undergo a 16 session exercise program for 2 months. Each session will last for 60minutes. The exercise program will be arranged in a group format with class size ranging from 6-8 per class. Subjects will be divided into experimental and control groups.
  Arms: Core stabilization exercise group

SUMMARY:
Objectives: To develop an exercise program for older adults with low back pain. And,to develop a clinical prediction rule that could identify a subgroup of people with NSLBP

Participants:

150 people aged between 40 to 80 with non-specific low back pain (NSLBP) for more than 6 months and is able to ambulate independently will be invited to join the study. People who had 1) previous spinal surgery; 2) LBP attributable to current pregnancy; 3) acute fracture, recent fall, tumour, or bone infection; and 4) experience of practising core-stability exercises in the past 6 months will be excluded. Study details will be explained to participants and written consent will be obtained prior the study. 75 participants will be randomized into the intervention group. Another 75 participants will be randomized into the waiting list control group.

Assessment Participants will undergo two comprehensive assessments before and after the training, which includes: Surface electromyogram (EMG) on the lumbar spine and abdominal muscle, Inertial measurement unit (IMU) sensor for trunk movement, clinical assessment including. Prone instability test.

Subjective assessments: Visual analogue scale score for pain, The Oswestry Low Back Pain Disability Questionnaire and Roland-Morris Disability Questionnaire.

Intervention - 16 session structured exercise program All participants will undergo a 16 session exercise program for 2 months. Each session will last for 60minutes. The exercise program will be arranged in a group format with class size ranging from 6 - 8 per class Subjects will be divided into experimental and control groups. Participants in the control group will not receive exercise training at first but were evaluated at the same time as participants in the experimental group. The participant in the control group completed the exercise training after the post-assessment.

DETAILED DESCRIPTION:
People with non-specific low back pain (NSLBP) demonstrate diversified clinical signs and symptoms. It is because the cause of NSLBP is multifaceted. Due to the varied pathophysiology and clinical behavior, the 'one-suit-all' approach of physiotherapy treatment prescription for people with NSLBP is usually less effective in reducing pain and improving daily function.

Research on identifying subgroups of patients with NSLBP who would benefit from physiotherapy interventions could provide clinicians evidence-based guidelines and enhance the cost-effectiveness of health care service. Earlier research showed that people with NSLBP demonstrated a delay in core muscle activation and general wasting of the trunk and core muscle. These pathological changes support the use of core stability training (e.g., Pilates exercise) to manage people with NSLBP. However, effectiveness of core stability training have not been studied extensively in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 1）people aged between 40 to 80 with non-specific low back pain (NSLBP) for more than 6 months ；2）people is able to ambulate independently

Exclusion Criteria:

* 1) previous spinal surgery; 2) LBP attributable to current pregnancy; 3) acute fracture, recent fall, tumour, or bone infection; and 4) experience of practising core-stability exercises in the past 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Low Back Pain Disability Questionnaire | pre-intervention session (T1)
  is a widely used questionnaire designed to assess the level of disability and functional impairment in individuals with lower back pain. The questionnaire consists of 10 sections, each focusing on a different aspect of daily living that might be affected by back pain, such as personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, and traveling.
  Each section is scored on a scale of 0 to 5, with higher scores indicating greater disability. The scores for all sections are then summed and converted to a percentage, which can range from 0% (no disability) to 100% (maximum disability).
The Oswestry Low Back Pain Disability Questionnaire | post-intervention (8 weeks after start of intervention;T2)
  is a widely used questionnaire designed to assess the level of disability and functional impairment in individuals with lower back pain. The questionnaire consists of 10 sections, each focusing on a different aspect of daily living that might be affected by back pain, such as personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, and traveling.
  Each section is scored on a scale of 0 to 5, with higher scores indicating greater disability. The scores for all sections are then summed and converted to a percentage, which can range from 0% (no disability) to 100% (maximum disability).

SECONDARY OUTCOMES:
Visual analogue scale (VAS) score for pain | pre-intervention session (T1)
  The Visual Analogue Scale (VAS) is a tool commonly used to measure a person's pain intensity. The scale typically consists of a 10cm horizontal line. Anchored by two verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most often anchored by "No Pain" at one end and "Worst Imaginable Pain" at the other.
  Patients are asked to mark a point along the line that represents their current level of pain.
Visual analogue scale (VAS) score for pain | post-intervention (8 weeks after start of intervention;T2)
  The Visual Analogue Scale (VAS) is a tool commonly used to measure a person's pain intensity. The scale typically consists of a 10cm horizontal line. Anchored by two verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most often anchored by "No Pain" at one end and "Worst Imaginable Pain" at the other.
  Patients are asked to mark a point along the line that represents their current level of pain.
Fear-Avoidance Belief Questionnaire | pre-intervention session (T1)
  Participants finish the questionnaire with the help of investigators to assess how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability.
  The scale score range from 0 - 96, a higher score indicates a higher level of fear avoidance beliefs.
Fear-Avoidance Belief Questionnaire | post-intervention (8 weeks after start of intervention;T2)
  Participants finish the questionnaire with the help of investigators to assess how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability.
  The scale score range from 0 - 96, a higher score indicates a higher level of fear avoidance beliefs.
Surface EMG | pre-intervention session (T1)
  EMG-sensors attached to the skin overlying the erector spinae at the T4 vertebrae (approximately 2-3 cm from the midline of the back) on both sides.
Surface EMG | post-intervention (8 weeks after start of intervention;T2)
  EMG-sensors attached to the skin overlying the erector spinae at the T4 vertebrae (approximately 2-3 cm from the midline of the back) on both sides.
IMU-sensor | pre-intervention session (T1)
  IMU-sensors attached to the skin overlying the erector spinae at the T3 and L1 vertebrae(approximately 3-4 cm from the midline of the back), Pelvis(S2) and femur. IMU-sensors were positioned unilaterally on the right side.
IMU-sensor | post-intervention (8 weeks after start of intervention;T2)
  IMU-sensors attached to the skin overlying the erector spinae at the T3 and L1 vertebrae(approximately 3-4 cm from the midline of the back), Pelvis(S2) and femur. IMU-sensors were positioned unilaterally on the right side.
Prone instability test | pre-intervention session (T1)
  Participants will assume a face-down position on a bench, allowing their legs to dangle off the edge so that their feet touch the ground. Manual pressure will then be applied on various lumbar spine segments to induce pain. If pain occurs, participants then raise their legs off the ground before the application of back-to-front pressure is repeated. A reduction in pain when lifting the legs indicates the ability to actively stabilize the spine, signifying a positive test result. In such cases, a stability-focused exercise regimen would be appropriate for the individual.
Prone instability test | post-intervention (8 weeks after start of intervention;T2)
  Participants will assume a face-down position on a bench, allowing their legs to dangle off the edge so that their feet touch the ground. Manual pressure will then be applied on various lumbar spine segments to induce pain. If pain occurs, participants then raise their legs off the ground before the application of back-to-front pressure is repeated. A reduction in pain when lifting the legs indicates the ability to actively stabilize the spine, signifying a positive test result. In such cases, a stability-focused exercise regimen would be appropriate for the individual.
straight leg raise (SLR) | pre-intervention session (T1)
  The Straight Leg Raise (SLR) test is a commonly used diagnostic procedure to evaluate for the presence of lumbar radiculopathy, often caused by a herniated disc. During the test, the patient lies flat on their back on an examination table. The examiner then lifts one of the patient's straightened legs by the ankle, keeping the knee extended.
straight leg raise (SLR) | post-intervention (8 weeks after start of intervention;T2)
  The Straight Leg Raise (SLR) test is a commonly used diagnostic procedure to evaluate for the presence of lumbar radiculopathy, often caused by a herniated disc. During the test, the patient lies flat on their back on an examination table. The examiner then lifts one of the patient's straightened legs by the ankle, keeping the knee extended
internal rotation range of motion | pre-intervention session (T1)
  When the knee is in a position of flexion between 30 and 90 degrees, there are approximately 45 degrees external and 25 degrees internal rotation. Rotatory motion decreases with further extension and, at 5 degrees of flexion, the knee has 23 degrees external and 10 degrees internal rotation.
internal rotation range of motion | post-intervention (8 weeks after start of intervention;T2)
  When the knee is in a position of flexion between 30 and 90 degrees, there are approximately 45 degrees external and 25 degrees internal rotation. Rotatory motion decreases with further extension and, at 5 degrees of flexion, the knee has 23 degrees external and 10 degrees internal rotation.
FABER test | pre-intervention session (T1)
  The FABER test is used to identify the presence of hip pathology by attempting to reproduce pain in the hip, lumbar spine or sacroiliac region. The test is a passive screening tool for musculoskeletal pathologies, such as hip, lumbar spine, or sacroiliac joint dysfunction, or an iliopsoas spasm.
FABER test | post-intervention (8 weeks after start of intervention;T2)
  The FABER test is used to identify the presence of hip pathology by attempting to reproduce pain in the hip, lumbar spine or sacroiliac region. The test is a passive screening tool for musculoskeletal pathologies, such as hip, lumbar spine, or sacroiliac joint dysfunction, or an iliopsoas spasm.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JH, Hoshino Y, Nakamura K, Kariya Y, Saita K, Ito K. Trunk muscle weakness as a risk factor for low back pain. A 5-year prospective study. Spine (Phila Pa 1976). 1999 Jan 1;24(1):54-7. doi: 10.1097/00007632-199901010-00013. PMID 9921591
- [Background] Kato S, Murakami H, Demura S, Yoshioka K, Shinmura K, Yokogawa N, Igarashi T, Yonezawa N, Shimizu T, Tsuchiya H. Abdominal trunk muscle weakness and its association with chronic low back pain and risk of falling in older women. BMC Musculoskelet Disord. 2019 Jun 3;20(1):273. doi: 10.1186/s12891-019-2655-4. PMID 31159812
- [Background] Arendt-Nielsen L, Graven-Nielsen T, Svarrer H, Svensson P. The influence of low back pain on muscle activity and coordination during gait: a clinical and experimental study. Pain. 1996 Feb;64(2):231-240. doi: 10.1016/0304-3959(95)00115-8. PMID 8740599
- [Background] Lamoth CJ, Meijer OG, Daffertshofer A, Wuisman PI, Beek PJ. Effects of chronic low back pain on trunk coordination and back muscle activity during walking: changes in motor control. Eur Spine J. 2006 Jan;15(1):23-40. doi: 10.1007/s00586-004-0825-y. Epub 2005 Apr 29. PMID 15864670
- [Background] Walter BA, Mageswaran P, Mo X, Boulter DJ, Mashaly H, Nguyen XV, Prevedello LM, Thoman W, Raterman BD, Kalra P, Mendel E, Marras WS, Kolipaka A. MR Elastography-derived Stiffness: A Biomarker for Intervertebral Disc Degeneration. Radiology. 2017 Oct;285(1):167-175. doi: 10.1148/radiol.2017162287. Epub 2017 May 4. PMID 28471737
- [Background] Roussel NA, Nijs J, Meeus M, Mylius V, Fayt C, Oostendorp R. Central sensitization and altered central pain processing in chronic low back pain: fact or myth? Clin J Pain. 2013 Jul;29(7):625-38. doi: 10.1097/AJP.0b013e31826f9a71. PMID 23739534
- [Background] Nakamura M, Nishiwaki Y, Sumitani M, Ushida T, Yamashita T, Konno S, Taguchi T, Toyama Y. Investigation of chronic musculoskeletal pain (third report): with special reference to the importance of neuropathic pain and psychogenic pain. J Orthop Sci. 2014 Jul;19(4):667-75. doi: 10.1007/s00776-014-0567-6. Epub 2014 Apr 16. PMID 24737064
- [Background] Assendelft WJ, Morton SC, Yu EI, Suttorp MJ, Shekelle PG. Spinal manipulative therapy for low back pain. A meta-analysis of effectiveness relative to other therapies. Ann Intern Med. 2003 Jun 3;138(11):871-81. doi: 10.7326/0003-4819-138-11-200306030-00008. PMID 12779297
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Fritz JM, Lindsay W, Matheson JW, Brennan GP, Hunter SJ, Moffit SD, Swalberg A, Rodriquez B. Is there a subgroup of patients with low back pain likely to benefit from mechanical traction? Results of a randomized clinical trial and subgrouping analysis. Spine (Phila Pa 1976). 2007 Dec 15;32(26):E793-800. doi: 10.1097/BRS.0b013e31815d001a. PMID 18091473
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Cooper RG, St Clair Forbes W, Jayson MI. Radiographic demonstration of paraspinal muscle wasting in patients with chronic low back pain. Br J Rheumatol. 1992 Jun;31(6):389-94. doi: 10.1093/rheumatology/31.6.389. PMID 1534505
- [Background] Danneels LA, Vanderstraeten GG, Cambier DC, Witvrouw EE, De Cuyper HJ. CT imaging of trunk muscles in chronic low back pain patients and healthy control subjects. Eur Spine J. 2000 Aug;9(4):266-72. doi: 10.1007/s005860000190. PMID 11261613
- [Background] Ravenna MM, Hoffman SL, Van Dillen LR. Low interrater reliability of examiners performing the prone instability test: a clinical test for lumbar shear instability. Arch Phys Med Rehabil. 2011 Jun;92(6):913-9. doi: 10.1016/j.apmr.2010.12.042. PMID 21621668
- [Background] Luomajoki H, Kool J, de Bruin ED, Airaksinen O. Reliability of movement control tests in the lumbar spine. BMC Musculoskelet Disord. 2007 Sep 12;8:90. doi: 10.1186/1471-2474-8-90. PMID 17850669
- [Background] Lue YJ, Hsieh CL, Huang MH, Lin GT, Lu YM. Development of a Chinese version of the Oswestry Disability Index version 2.1. Spine (Phila Pa 1976). 2008 Oct 1;33(21):2354-60. doi: 10.1097/BRS.0b013e31818018d8. PMID 18827702
- [Background] Aladro-Gonzalvo AR, Araya-Vargas GA, Machado-Diaz M, Salazar-Rojas W. Pilates-based exercise for persistent, non-specific low back pain and associated functional disability: a meta-analysis with meta-regression. J Bodyw Mov Ther. 2013 Jan;17(1):125-36. doi: 10.1016/j.jbmt.2012.08.003. Epub 2012 Sep 16. PMID 23294694